CLINICAL TRIAL: NCT02286310
Title: Effect of Exercise Programs on 3-dimensional Scapular Kinematics, Disability and Pain in Subjects With Shoulder Impingement
Brief Title: Effect of Exercise Programs on 3-dimensional Scapular Kinematics, Disability and Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Elif Turgut, Research Assistant, Physiotherapy, MSc, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO14-189
Record Dates: First submitted 2014-11-02; First posted 2014-11-07 (Estimated); Last update posted 2014-11-10 (Estimated); Status verified 2014-11

CONDITIONS: Shoulder Impingement Syndrome
Keywords: Exercise; Kinematics
MeSH Terms: conditions — Shoulder Impingement Syndrome; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group A (Experimental): Kinetic Chain Exercises
  Interventions: Other: Kinetic Chain Exercises
- Group B (Active Comparator): Traditional Exercises
  Interventions: Other: Traditional Exercises

INTERVENTIONS:
Other: Kinetic Chain Exercises — Exercises include kinetic chain segments.
  Arms: Group A
Other: Traditional Exercises — Stretching, strengthening exercises.
  Arms: Group B

SUMMARY:
The aim of this study is to investigate the effect of exercise program on 3-dimensional scapular kinematics, disability and pain on shoulder impingement with scapular dyskinesia.

ELIGIBILITY:
Inclusion Criteria:

* Subacromial impingement with scapular dyskinesia

Exclusion Criteria:

* Additional muscular and skeletal or systemic diseases

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2014-02; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
3-Dimensional Scapular Kinematics measured by electromagnetic tracking system | Change from Baseline in Angular Data at 1 year
  Scapular rotations and orientations in degrees

SECONDARY OUTCOMES:
Pain and Disability Status measured by Shoulder Pain and Disability Index (SPADI) | Change from Baseline in Scor at 1 year
  Scoring with patient-reported outcome measure
Pain Severity measured by Visual Analogue Scale (in millimeters) | Change from Baseline in Pain Severity at 1 year
  Scale is in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Gul Baltaci, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Derived] Turgut E, Duzgun I, Baltaci G. Effects of Scapular Stabilization Exercise Training on Scapular Kinematics, Disability, and Pain in Subacromial Impingement: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2017 Oct;98(10):1915-1923.e3. doi: 10.1016/j.apmr.2017.05.023. Epub 2017 Jun 24. PMID 28652066